## Değerli Katılımcı,

Bu çalışmada, tek kanallı elektroensefalografi ve fotopletismografi sensörlerininin kombinasyonunu içeren bir cihaz ve bir yazılım yardımı ile temel uyku evreleri, kalp atım hızı, kalp atım hızı değişkenliği ve oksijen satürasyonu çıktılarının hesaplanmaları yapılacaktır. Hedeflediğimiz çıktıların daha önce güvenilirlik geçerlilikleri yapılmış cihazlar ile karşılaştırmalarının yapılması bu çalışmanın amacıdır.

Bunun için hali hazırda gönüllü olarak uyku testi yaptırmak üzere yatmış olduğunuz İstanbul Tıp Fakültesi Uyku Bozukluk merkezinde, polisomnografi cihazına ek olarak alın bölgenize (EEG ve ışık sensörü) ve el bileğinize (ışık sensörü) sensör takılacaktır. Bu sensör, size zarar vermeyecek, canınızı yakmayacak ve dokunuzda herhangi bir hassasiyete yol açmayacaktır. Sensörler genişlik ve yükseklik olarak çok yer kaplamamaktadır ve kablosuz çalışmaktadır. Bu size ekstra kablo sorunu çıkarmadığımızı göstermektedir.

Çalışmamızın sonunda, karşılaştırmalarını yapacağımız parametreler öncesinde belirlediğimiz sınır değerler ile uyuşursa (performans başarısı yakalanırsa), kendi ortamınızda uykunuzu, kalp atım hızı, kalp atım hızı değişkenliğinizi ve oksijen satürasyonunuzu takip edebileceğiniz bir cihaz kullanma ihtimaline sahip olacaksınız. Bu cihaz yardımı ile birçok vücudun birçok bölgesine yerleştirilen elektrot ve kablodan kurtulunacak ve ölçüm konforu artacaktır.

Çalışmamız süresince hastane doktorlarından olan ve Marmara Üniversitesinde görev yapan her zaman teknik destek, sorularınız yanıtlanması ve sonuçların yorumlanması kısmı için iletişime açık olacaktır.

Çalışma kapmasında, katıldığınız uyku ölçümde ilave olarak iki sensör takılmasının dışında yapmanızı istediğimiz hiçbir eylem ve bununla beraber gelen bir sorumluluk bulunmamaktadır.

Yukarıda açıkça tanımlanan çalışmanın ne amaçla, kimler tarafından ve nasıl gerçekleştirileceği anlayabileceğim bir ifade ile bana anlatıldı.

Çalışma sırasında hekim ile aramda kalması gereken bana ait bilgilerin gizliliğine bu araştırma sırasında da büyük özen ve saygı ile yaklaşılacağına inanıyorum. Araştırma sonuçlarının eğitim ve bilimsel amaçlarla kullanımı sırasında kişisel bilgilerimin ihtimamla korunacağı konusunda bana yeterli güven verildi.

Bu çalışmadan elde edilen bilgilerin bana ve başka insanlara sağlayacağı yararlar bana anlatıldı.

Çalışmaya hiçbir baskı ve zorlama altında olmaksızın gönüllü olarak katılıyorum.

Sorumlu araştırmacıya haber vermek kaydıyla, hiçbir gerekçe göstermeksizin istediğim anda bu çalışmadan çekilebileceğimin bilincindeyim.

Çalışmanın yürütücüsü olan araştırmacı veya destekleyen kuruluş, çalışma programının gereklerini yerine getirmedeki ihmalim nedeniyle, benim onayımı almadan beni çalışma kapsamından çıkarabilir.

Çalışmanın sonuçları bilimsel toplantılar ya da yayınlarda sunulabilir. Ancak, bu tür durumlarda kimliğim kesin olarak gizli tutulacaktır.

Aklıma gelen bütün soruları sorma olanağı tanındı ve sorularıma cevaplar aldım. Bu koşullarla, söz konusu araştırmaya hiçbir baskı ve zorlama olmaksızın gönüllü olarak katılmayı kabul ediyorum.

Sayın tarafından İstanbul Tıp Fakültesi Uyku Bozuklukları Merkezinde hali hazırda yaptıracağım uyku testi sırasında böyle bir çalışmanın yürütülebileceği ve bu çalışmada gönüllü katılımcı olabileceğim söylendi ve çalışmaya davet edildim.

Araştırma sırasında bir sağlık sorunu ile karşılaştığımda; herhangi bir saatte, telefon numaralarından, İstanbul Tıp Fakültesi/Topkapı, Turgut Özal Millet Cd No:118 D:118, 34093 Fatih/İstanbul ve Spor Bilimleri Fakültesi, Spor Sağlık Bilimleri Anabilim dalı Göksu Mah. Cuma Yolu Cad. No:1 Marmara Yerleşkesi PK. 34815- Beykoz/İstanbul adreslerinden arayabileceğimi biliyorum.

Çalışmaya katılmam konusunda zorlayıcı bir davranışla karşılaşmış değilim. Eğer katılmayı reddedersem, bu durumun tıbbi bakımıma ve hekim ile olan ilişkime herhangi bir zarar getirmeyeceğini de biliyorum.

Bana yapılan tüm açıklamaları ayrıntılarıyla anlamış bulunmaktayım. Kendi başıma belli bir düşünme süresi sonunda isimli çalışmaya "katılımcı" (denek) olarak yer alma kararını aldım. Bu konuda yapılan daveti gönüllülük içerisinde kabul ediyorum. İmzalamış bulunduğum bu form kâğıdının bir kopyası bana verilecektir.

## GÖNÜLLÜ ONAY FORMU

Yukarıda gönüllüye araştırmadan önce verilmesi gereken bilgileri gösteren metni okudum. Bunlar hakkında bana yazılı ve sözlü açıklamalar yapıldı. Bu koşullarla söz konusu klinik araştırmaya kendi rızamla hiçbir baskı ve zorlama olmaksızın katılmayı kabul ediyorum.

Gönüllünün Adı-soyadı, İmzası, Adresi

Velayet veya vesayet altında bulunanlar için veli veya vasinin adı-soyadı, imzası, adresi

Açıklamaları yapan araştırmacının adı-soyadı, imzası

Rıza alma işlemine başından sonuna kadar tanıklık eden kuruluş görevlisinin adı-soyadı, imzası, görevi